CLINICAL TRIAL: NCT02717832
Title: Protection Against Insulin Resistance in Obesity
Acronym: PAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science and Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00111275
Record Dates: First submitted 2016-03-07; First posted 2016-03-24 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Sensitivity (Experimental)
  Interventions: Drug: hyperinsulinemic-euglycemic clamp

INTERVENTIONS:
Drug: hyperinsulinemic-euglycemic clamp

SUMMARY:
The overall goal of this project is to identify factors that "protect" some obese adults from becoming insulin resistant. Identifying mechanisms that help protect some obese adults from developing insulin resistance could lead to novel, targeted therapeutic and/or preventative strategies for obese adults who are insulin resistant.

DETAILED DESCRIPTION:
SCREENING PROCEDURES Participants will undergo a battery of initial screening tests including: a detailed health history and physical examination, a physical activity questionnaire, and a body composition assessment. All women will undergo a urine pregnancy test.

GENERAL STUDY DESIGN To avoid potential confounding hormonal effects, all women will be studied in the early follicular phase of their menstrual cycle. Subjects will be advised of what they should be eating in the 3 days leading up to their hospital visit to maintain their weight. Subjects will also complete a three day food journal before their hospital visit. The day prior to the study trial admission, subjects will need to eat pre-prepared standardized meals for breakfast, lunch, dinner and an evening snack that the study team has given them.

Subjects will be admitted to the Michigan Clinical Research Unit (MCRU) in the morning after a 12-hour, overnight fast. After arrival, subjects will rest quietly in their room for about 30 minutes. The study team will then measure subjects resting metabolic rate for about 20 minutes. After this test, an intravenous (IV) catheter will be placed for infusions and a second IV will be placed in vein of the opposite arm for blood sampling.

After the IV placement, the study team will begin a tracer-labeled glucose, or "sugar," infusion. The study team will then remove a small sample of muscle from the subjects thigh. This muscle biopsy procedure involves numbing a nickel-sized portion of the skin of the thigh with a local anesthetic, making a small incision (1/4 inch), and removing a small piece of muscle (approximately the size of 2-3 grains of rice). The incision will then be closed with a piece of sterile tape. The study team will also obtain a small sample of fat tissue from the area just underneath the skin near the belly button. This procedure involves numbing a small region of skin near the belly button with a local anesthetic, using a needle a small amount of fat tissue is removed from underneath the skin. During the procedure subjects will feel some pinching and pulling, but it should not be very painful. The injury resulting from the muscle and fat tissue biopsies is rather minor. Subjects will likely have some bruising and mild soreness, but it should not prevent them from performing their general daily activities.

Approximately 2.5 hours after admission, the study team will begin the tracer-labeled fat infusion. The tracer-labeled fats the study team are infusing occur naturally in the body. By injecting a slightly greater amount of this substance than what is already in the body the study team will be able to measure the rate of fat breakdown and fat burning. After about 50 minutes of the infusion, three blood samples will be obtained in 5 min intervals.

After, the study team will begin a hyperinsulinemic-euglycemic clamp procedure (a procedure to measure the body's sensitivity to insulin). During this procedure the study team will infuse insulin and glucose through the IV and will collect blood samples every 5 minutes for the duration of the procedure to monitor the subjects blood glucose and blood insulin concentrations. This procedure is designed to last 2 hours. The study team will change the infusion rate of glucose accordingly to ensure that the subjects blood sugar is maintained at a healthy/normal level. The study team will also infuse a small amount of potassium to make sure potassium concentrations remain at healthy/normal levels. About 30 minutes after starting this procedure to measure the body's sensitivity to insulin, the study team will collect another sample of muscle from the thigh and fat tissue from the area just underneath the skin near the belly button. After completing the hyperinsulinemic-euglycemic clamp procedure, subjects will be provided a meal, and the study team will continue to monitor the subjects blood glucose concentration until stable.

When the subjects vital signs are stable, the study team will also measure percent body fat using a Dual Energy X-ray Absorptiometry (DEXA) and intra-abdominal fat by Magnetic resonance imaging (MRI). When the DEXA scan and MRI tests have been completed, subjects will be discharged from the hospital. Depending on scheduling, however, the DEXA scan and MRI tests may be performed on a separate occasion from the study trial admission.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [BMI]: 30-40 kg/m2
* Age: 18-45 years
* All women must be pre-menopausal
* Non-exerciser: no regularly planned exercise/physical activity

Exclusion Criteria:

* Weight instability ≥ ±3kg ≥ 6 months
* Medications known to affect lipid and/or glucose metabolism
* Pregnancy or actively breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Sensitivity: hyperinsulinemic-euglycemic clamp
Period: Overall Study
Arm/Group | Insulin Sensitivity
Started | 20
Completed | 17
Not Completed | 3
Not completed — Inability to place IV | 3

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Sensitivity
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity
Time Frame: baseline (this cross-sectional study involves only one insulin sensitivity measurement in a single visit for each participant)
Population: BMI: 30-40 kg/m2; waist circumference: 88-98cm for women and 100-110cm for men), age: 18-45 years old), weight stable (±3kg for ≥ 6 months), No medications known to affect lipid or glucose metabolism. No evidence and/or history of cardiovascular or metabolic diseases All women were pre-menopausal with regularly occurring menses.
Measure: Mean (Standard Deviation); unit: nmol/kg FFM/min /(µU/mL Insulin)
Groups:
- Low Insulin Sensitivity Group: Adults with obesity with a rate of glucose disappearance from plasma (Rd Glucose) < 400 nmol/kg fat free mass/min/(uU/ml Insulin)
- High Insulin Sensitivity Group: Adults with obesity with a rate of glucose disappearance from plasma (Rd Glucose) >550 nmol/kg fat free mass/min/(uU/ml Insulin)
Arm/Group | Low Insulin Sensitivity Group | High Insulin Sensitivity Group
Number analyzed (Participants) | 10 | 7
nmol/kg FFM/min /(µU/mL Insulin) | 273 (54) | 817 (257)

2. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate was measured using a metabolic cart (to measure VO2 and VCO2) in the morning after an overnight fast
Time Frame: baseline (this cross-sectional study involves only one Resting Metabolic Rate measurement in a single visit for each participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | Low Insulin Sensitivity Group | High Insulin Sensitivity Group
Number analyzed (Participants) | 8 | 6
kcals/day | 1509 (237) | 1325 (198)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Insulin Sensitivity
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT02717832/Prot_SAP_000.pdf